CLINICAL TRIAL: NCT05856084
Title: A Phase II, Single Center, Randomized, Blind, Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Recombinant Herpes Zoster Vaccine (CHO Cells) in Healthy Subjects Aged 30 Years and Above
Brief Title: Immunogenicity and Safety of Recombinant Herpes Zoster Vaccine (CHO Cells) in Healthy Subjects Aged 30 Years and Above
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT-100-002
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Low dose vaccine group in adults aged 30 to 49 years (Experimental): Participants aged 30 to 49 years will be vaccinated with 2 doses of low dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low dose Recombinant Herpes Zoster Vaccine (CHO cells)
- High dose vaccine group in adults aged 30 to 49 years (Experimental): Participants aged 30 to 49 years will be vaccinated with 2 doses of high dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High dose Recombinant Herpes Zoster Vaccine (CHO cells)
- Placebo group in adults aged 30 to 49 years (Placebo Comparator): Participants aged 30 to 49 years will be vaccinated with 2 doses of placebo on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Placebo
- Low dose vaccine group in adults aged 50 years and older (Experimental): Participants aged 50 years and older will be vaccinated with 2 doses of low dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low dose Recombinant Herpes Zoster Vaccine (CHO cells)
- High dose vaccine group in adults aged 50 years and older (Experimental): Participants aged 50 years and older will be vaccinated with 2 doses of high dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High dose Recombinant Herpes Zoster Vaccine (CHO cells)
- Shingrix® group in adults aged 50 years and older (Active Comparator): Participants aged 50 years and older will be vaccinated with 2 doses of Shingrix® on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Positive control
- Placebo group in adults aged 50 years and older (Placebo Comparator): Participants aged 50 years and older will be vaccinated with 2 doses of placebo on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose Recombinant Herpes Zoster Vaccine (CHO cells) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with low dose MA105.
  Arms: Low dose vaccine group in adults aged 30 to 49 years; Low dose vaccine group in adults aged 50 years and older
Biological: High dose Recombinant Herpes Zoster Vaccine (CHO cells) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with high dose MA105.
  Arms: High dose vaccine group in adults aged 30 to 49 years; High dose vaccine group in adults aged 50 years and older
Biological: Positive control — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with AS01B.
  Other Names: Shingrix®
  Arms: Shingrix® group in adults aged 50 years and older
Biological: Placebo — 0.5 mL per dose, containing 4.5 mg sodium chloride.
  Other Names: Normal Saline for injection
  Arms: Placebo group in adults aged 30 to 49 years; Placebo group in adults aged 50 years and older

SUMMARY:
The purposes of the study are to evaluate the immunogenicity and safety of different dose levels of recombinant herpes zoster vaccine (CHO Cells) with 2 doses at 2-month intervals in healthy subjects aged 30 years and older.

DETAILED DESCRIPTION:
The clinical trial will be a single-center, randomized, blind, controlled study in which two dose levels of vaccine will be tested in healthy adults aged 30 to 49 years and 50 years and older. A total of 924 participants will be enrolled, including 396 participants aged 30 to 49 years and 528 participants aged 50 years and older. Participants aged 30 to 49 years will be randomized into three subgroups (low dose vaccine group, high dose vaccine group and placebo group) in a 1:1:1 ratio. Participants aged 50 years and older will be randomized into four subgroups (low dose vaccine group, high dose vaccine group, Shingrix® group and placebo group) in a 1:1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent residents aged 30 years and above;
2. Subjects voluntarily agree to participate in the study and signed an informed consent;
3. Be able to participate in all scheduled visits and comply with the protocol requirements.

Exclusion Criteria:

1. Axillary temperature>37.0℃;
2. History of herpes zoster within 5 years before vaccination;
3. Prior vaccination with chickenpox vaccine or herpes zoster vaccine;
4. Female participant who is pregnant ( urine pregnancy test was positive) or breastfeeding, or has pregnancy plans within 1 year after the last vaccination;
5. Receipt of live vaccine within 28 days, or any other vaccine within 14 days prior to vaccination;
6. Receipt of immunoglobulin or intravenous immunoglobulin within 3 months before vaccination;
7. Acute diseases or acute exacerbation of chronic disease within 3 days before vaccination;
8. A known allergy to any components of the study vaccine (especially allergic to aminoglycoside antibiotics), or history of severe allergy to any previous vaccination;
9. History of convulsions, epilepsy, encephalopathy (such as congenital brain dysplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral infarction, brain infection disease, nerve tissue damage caused by chemical drug poisoning, etc.) or mental illness and family history;
10. Asplenia or functional asplenia, or splenectomy caused by any condition;
11. Primary or secondary impairment of immune function or diagnosed congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases;
12. Receipt of immunosuppressive therapy within 3 months before vaccination (such as long-term use of systemic glucocorticoid ≥14 days, dose ≥2mg/kg/day or ≥20mg/day prednisone or equivalent dose), but inhaled, intra-articular and topical steroids are acceptable;
13. Severe cardiovascular disease(eg. Pulmonary heart disease, Pulmonary Edema); Severe liver or kidney disease; or diabetes with complication;
14. History of thrombocytopenia or other coagulation disorders, which may cause intramuscular injection contraindications;
15. Abnormal blood pressure during physical examination before vaccination (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mmHg);
16. Current or history of alcohol and/or drug abuse;
17. Any condition that, in the opinion the investigator, may affect the safety of the subject or the evaluation of the study results.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2023-05-07 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean concentration (GMC) of anti-gE antibody | Month 1 after the last vaccination
  Measured by ELISA.
Seropositivity rate of anti-gE antibody | Month 1 after the last vaccination
  The seropositivity rate is defined as the percentage of seropositive subjects. A seronegative subject is a subject whose antibody concentration is below the cut-off value. A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value.
Seroresponse rate of anti-gE antibody | Month 1 after the last vaccination
  The seroresponse rate is defined as the percentage of subjects who have at least a: 4-fold increase in the antibody concentration as compared to the pre vaccination antibody concentration, for subjects who are seropositive at baseline, OR, 4-fold increase in the antibody concentration as compared to the antibody concentration cut-off value for seropositivity, for subjects who are seronegative at baseline.
Geometric Mean Fold Rise (GMFR) of anti-gE antibody concentration | Month 1 after the last vaccination
  The antibody concentration at month 1 after the last vaccination compared with that at baseline (Day 0).
Four-fold increase rate of anti-gE antibody concentration | Month 1 after the last vaccination
  The antibody concentration at month 1 after the last vaccination compared with that at baseline (Day 0).
Cell-Mediated Immunity (CMI) response | Month 1 after the last vaccination
  CMI response is defined as the frequency of CD4+ T cells producing at least 2 activation markers (IFN-γ, IL-2, TNF-α and/or CD40L) upon in vitro stimulation by gE peptide pools.
Vaccine Response Rate (VRR) | Month 1 after the last vaccination
  VRR is defined as the percentage of participants with T-cell frequencies are ≥Cut-off value, for participants with T-cell frequencies<Cut-off at baseline, OR, at least a 2-fold increase as compared to baseline for participants with T-cell frequencies ≥Cut-off value at baseline.
The incidence and severity of adverse events | Within 30 minutes after each vaccination
  Incidence and severity of adverse events within 30 minutes after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence and severity of adverse events | Within 7 days after each vaccination
  Incidence and severity of adverse events within 7 days after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence and severity of adverse events | Day 8 to 30 after each vaccination
  Incidence and severity of adverse events during Day 8 to 30 after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence and severity of adverse events | Within 30 days after each vaccination
  Incidence and severity of adverse events within 30 days after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.

SECONDARY OUTCOMES:
The incidence of Serious Adverse Events | From the first vaccination to 12 months after the last vaccination
  Incidence of Serious Adverse Events (SAEs) from the first vaccination to 12 months after the last vaccination.
Potential Immune-Mediated Diseases | From the first vaccination to 12 months after the last vaccination
  Incidence of Potential Immune-Mediated Diseases (pIMDs) from the first vaccination to 12 months after the last vaccination.
Geometric mean concentration (GMC) of anti-VZV antibody | Month 1 after the last vaccination
  measured by ELISA.
Seropositivity rate of anti-VZV antibody | Month 1 after the last vaccination
  The seropositivity rate is defined as the percentage of seropositive subjects. A seronegative subject is a subject whose antibody concentration is below the cut-off value. A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value.
Seroresponse rate of anti-VZV antibody | Month 1 after the last vaccination
  The seroresponse rate is defined as the percentage of subjects who have at least a: 4-fold increase in the antibody concentration as compared to the pre vaccination antibody concentration, for subjects who are seropositive at baseline, OR, 4-fold increase in the antibody concentration as compared to the antibody concentration cut-off value for seropositivity, for subjects who are seronegative at baseline.
Geometric Mean Fold Rise (GMFR) of anti-VZV antibody | Month 1 after the last vaccination
  The antibody concentration at month 1 after the last vaccination compared with that at baseline (Day 0).
Four-fold increase rate of anti-VZV antibody | Month 1 after the last vaccination
  The antibody concentration at month 1 after the last vaccination compared with that at baseline (Day 0).
Geometric mean concentration (GMC) of anti-gE antibody | At 6, 12 and 24 months after the last vaccination
  measured by ELISA.
Seropositivity rate of anti-gE antibody | At 6, 12 and 24 months after the last vaccination
  The seropositivity rate is defined as the percentage of seropositive subjects. A seronegative subject is a subject whose antibody concentration is below the cut-off value. A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value.
Geometric mean concentration (GMC) of anti-VZV antibody | At 6, 12 and 24 months after the last vaccination
  measured by ELISA.
Seropositivity rate of anti-VZV antibody | At 6, 12 and 24 months after the last vaccination
  The seropositivity rate is defined as the percentage of seropositive subjects. A seronegative subject is a subject whose antibody concentration is below the cut-off value. A seropositive subject is a subject whose antibody concentration is greater than or equal to the cut-off value.
Cell-Mediated Immunity (CMI) response | At 6, 12 and 24 months after the last vaccination
  CMI response is defined as the frequency of CD4+ T cells producing at least 2 activation markers (IFN-γ, IL 2, TNF-α and/or CD40L) upon in vitro stimulation by gE peptide pools.
Vaccine Response Rate (VRR) | At 6, 12 and 24 months after the last vaccination
  VRR is defined as the percentage of participants with T-cell frequencies are ≥Cut-off value, for participants with T-cell frequencies<Cut-off at baseline, OR, at least a 2-fold increase as compared to baseline for participants with T-cell frequencies ≥Cut-off value at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Yanjin Center for Disease Control and Prevention, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No